CLINICAL TRIAL: NCT02260973
Title: The Influence of PRN Omega-3 Nutritional Supplement on Visual Acuity Outcomes In Cases Undergoing Cataract Surgery: A Pilot Study.
Brief Title: The Influence of PRN Omega-3 Nutritional Supplement on Visual Acuity
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Physician Recommended Nutriceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PRN 20145
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Cataract, Dry Eye Disease
MeSH Terms: conditions — Cataract; Dry Eye Syndromes | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Omega-3 (Active Comparator): re esterified TG omega-3
  Interventions: Dietary Supplement: Omega-3 (Triglyceride form)
- Safflower Oil (Placebo Comparator): vegetable oil
  Interventions: Dietary Supplement: Omega-3 (Triglyceride form)

INTERVENTIONS:
Dietary Supplement: Omega-3 (Triglyceride form)

SUMMARY:
This is a randomized, masked, placebo controlled study to assess the effect on visual acuity, if any, of the PRN omega-3 nutritional supplement in subjects undergoing cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Presence of nuclear or cortical lens opacities in one/both eyes
* Physician diagnosis of age related cataract
* Good overall physical constitution
* All participants must be follow the same regimen for surgery related medications, both pre and post surgery. (Antibiotic, NSAID and Steroid eye drops)

Exclusion Criteria:

* Subjects requiring Premium IOLs/multifocal implants
* Advanced cataract
* Severe Age-Related Macular Degeneration Presence or history of Glaucoma
* Presence or history of Diabetes Mellitus
* Any Retinal pathology - retinal detachment, retinitis pigmentosa, diabetic retinopathy, etc
* Vision loss due to Central retinal artery occlusion or Central retinal vein occlusion
* Vision loss due to presence of large pituitary tumors or aneurysms
* Vision loss due to optic tract lesions
* Vision loss due to bleeding into aqueous or vitreous chamber
* Vision loss due to drug toxicity: Amiodarone, anti-tuberculosis drugs, hydroxychloroquine, tamoxifen
* Major cardiovascular or cerebral events in the past 12 months
* Allergy to fish oil or safflower oil
* Pregnancy or lactation at any time during the study
* Newly started or increased the dose of chronic systemic medication known to affect tear production including, but not limited to antihistamines, antidepressants, diuretics, corticosteroids or immunomodulators within 30 days of Screening or at any time during the study
* Participation in any other study involving an investigational drug or device within the past 30 days

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Williams, MD, Principal Investigator — Southern Eye Associates
Locations (2):
- United States (2):
  - Cincinnati Eye Institute, Lexington, Kentucky
  - Southern Eye Associates, Greenville, South Carolina